CLINICAL TRIAL: NCT04443673
Title: Controlled and Randomized Clinical Trial for Evaluating the Effect of a Supplement of Glycine as Adjuvant in the Treatment of COVID-19 Pneumonia in Patients Initiating Mechanical Ventilation
Brief Title: Glycine Supplement for Severe COVID-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An interim analysis showed no difference in major outcomes (n=35 glycine and n=24 control participants)
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Mario H. Vargas, Senior Researcher, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C40-20
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; SARS-CoV Infection; SARS (Severe Acute Respiratory Syndrome); SARS Pneumonia; ARDS, Human; Pneumonia, Viral
Keywords: Glycine; Aminoacetic Acid; Coronavirus Disease; COVID-19; Severe Acute Respiratory Syndrome; SARS
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome; Pneumonia, Viral | interventions — Glycine

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, two branches, clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycine (Experimental): Along with habitual treatment for their severe condition, participants will receive 0.5 g/kg/day glycine by nasogastric tube, divided in four equal doses in a day, since their enrollment and until they are weaned from mechanical ventilator or die.
  Interventions: Dietary Supplement: Glycine
- Control (No Intervention): Participants will receive the habitual treatment for their severe condition.

INTERVENTIONS:
Dietary Supplement: Glycine — Along with habitual treatment for their severe condition, participants will receive 0.5 g/kg/day glycine by nasogastric tube, divided in four equal doses in a day, since their enrollment and until they are weaned from mechanical ventilator or die.
  Arms: Glycine

SUMMARY:
This study will explore whether a daily supplement of glycine, a substance that has antiinflammatory, cytoprotective, and endothelium-protecting effects, can improve mortality, as well as clinical and biochemical parameters, in patients with severe COVID-19 who initiate mechanical ventilatory support.

DETAILED DESCRIPTION:
Patients with severe forms of COVID-19 often develop acute respiratory distress syndrome (ARDS) associated with high levels of proinflammatory cytokines and damage of lungs and other organs. A special feature in these patients is thrombotic events in the micro- and macro-vasculature. Owing to the lack of a specific and efficient treatment against COVID-19, lowering of this "cytokine storm" is a further proposed strategy.

Glycine is the major agonist of glycine receptors (GlyR), which are chloride channels that hyperpolarize cell membranes of inflammatory cells such as macrophages and neutrophils, turning them less sensitive to proinflammatory stimuli. In addition, glycine possesses a cytoprotective effect, improves endothelial function, and diminishes platelet aggregation.

In laboratory animals, in a rat model of endotoxic shock a 5% glycine-rich diet lowers mortality, reduces pulmonary neutrophilic inflammation and hepatic lesions, and avoids elevation of serum TNF-alpha. In animal models of ischemia-reperfusion injury, glycine protects the gut and lungs.

In in vitro studies, glycine diminishes the expression and release of TNF-alpha and IL-6 from adipose tissue, 3T3-L1 cells, and alveolar macrophages, probably through inhibition of phosphorylation of NF-kappaB. Finally, glycine diminishes platelet aggregation.

In human beings, glycine has been used for many years for the management of some ailments. In diabetic patients, oral glycine reduces glycosylated hemoglobin levels and serum TNF-alpha, and in patients with cystic fibrosis glycine improves the clinical and spirometric status, and tend to lower serum TNF-alpha, IL-6 and G-CSF.

Glycine is a white microcrystal powder soluble in water, with a sweet taste and relatively low cost.

This controlled, randomized, two-branches clinical trial will recruit participants of any sex, any age, with COVID-19 confirmed (or awaiting confirmation) by PCR, that are to initiate (or with <48 h of) mechanical ventilation. After obtaining an informed consent, participants will be randomly assigned to two branches: 1) Experimental group, n=41 participants, that along with habitual management for their condition will receive 0.5 g/kg/day glycine divided in four doses every 6 h through nasogastric tube. 2) Control group, n=41 participants that will only receive habitual management. Pregnant women and subjects already participating in another study protocol will be excluded, and those with voluntary discharge or referenced to another institution will be discarded.

Blood samples for measurements of serum cytokines (Bio-Plex Human Cytokine 17-Plex, Bio-Rad) will be obtained at the beginning of the study and every 7 days thereafter.

The major outcome will be mortality. Secondary outcomes will be diminution of number of days under mechanical ventilation and evolution of PaO2/FiO2, proinflammatory and metabolic biomarkers, Sequence Organ Failure Assessment (SOFA), and Acute Physiology and Chronic Health Evaluation II (APACHE II).

Routine test such as arterial blood gases, blood chemistry, blood count, coagulation test, and ECG will also be analyzed by using the weighted average in certain time-periods (probably 7-days periods).

Group comparisons will be carried out by means of Fisher exact/chi-square tests and Student's t-/Mann-Whitney U-tests. Feasibility of multivariate analysis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Any age.
* Any sex.
* With COVID-19 confirmed (or awaiting confirmation) by PCR.
* With a clinical decision of initiation of mechanical ventilation or with <48 h under mechanical ventilation.
* Informed consent signed by the participant's responsible.

Exclusion Criteria:

* Pregnant women.
* Already participating in another research protocol.

Elimination Criteria:

* Voluntary hospital discharge or referenced to another institution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of participants who die divided by number of subjects enrolled in the that study group.

SECONDARY OUTCOMES:
Days under mechanical ventilation | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of days spent under mechanical ventilation.
PaO2/FiO2 ratio | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Arterial pressure of oxygen divided by inspired fraction of oxygen.
Arterial plasma lactate | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Plasma concentration of lactate in arterial blood.
Serum IL-1β | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 1β.
Serum IL-2 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 2.
Serum IL-4 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 4.
Serum IL-5 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 5.
Serum IL-6 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 6.
Serum IL-7 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 7.
Serum IL-8 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 8.
Serum IL-10 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 10.
Serum IL-12 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 12 (p70).
Serum IL-13 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 13.
Serum IL-17 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interleukin 17A.
Serum G-CSF | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of granulocyte colony stimulating factor.
Serum GM-CSF | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of granulocyte monocyte colony stimulating factor.
Serum IFN-γ | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of interferon gamma.
Serum MCP-1 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of monocyte chemoattractant protein 1 (MCAF).
Serum MIP-1β | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of macrophage inflammatory protein 1β
Serum TNF-α | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of tumor necrosis factor alpha.
Serum creatinine | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of creatinine.
Serum alanine aminotransferase | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of alanine aminotransferase.
  .
Serum aspartate aminotransferase | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of aspartate aminotransferase.
  .
Serum alkaline phosphatase | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of alkaline phosphatase.
Serum total bilirubin | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of total bilirubin.
Serum unconjugated bilirubin | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of unconjugated bilirubin.
Serum conjugated bilirubin | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of conjugated bilirubin
Serum C reactive protein | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of C reactive protein.
Hemoglobin | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Blood concentration of hemoglobin.
Total leukocytes | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of white blood cells per µl blood.
Neutrophils | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of neutrophils per µl blood.
Lymphocytes | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of lymphocytes per µl blood.
Monocytes | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of monocytes per µl blood.
Eosinophils | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of eosinophils per µl blood.
Basophils | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of basophils per µl blood.
Platelets | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Number of platelets per µl blood.
Prothrombin time | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Time that blood takes to clot.
Serum PAI-1 | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Serum concentration of plasminogen activator inhibitor 1 (PAI-1).
SOFA score | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Sequence Organ Failure Assessment (SOFA) score, composed by assessment of PaO2/FiO2 ratio, Glasgow coma scale, mean arterial pressure, bilirubin, and platelets.
APACHE II score | From date of enrollment and until the date of weaning from ventilator or death, whichever came first, assessed up to 12 months.
  Acute Physiology And Chronic Health Evaluation II (APACHE II) score, composed by assessment of AaDO2 or PaO2, temperature, mean arterial pressure, pH arterial, heart rate, respiratory rate, sodium, potassium, creatinine, hematocrit, white blood cell count, Glasgow coma scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mario H Vargas, MSc, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared on a reasonable basis and after authorization from the Instituto Nacional de Enfermedades Respiratorias' IRB.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From publication of results in a scientific journal onward.
Access Criteria: Reasonable request by E-mail (mhvargasb@yahoo.com.mx)

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Yang Y, Shen C, Li J, Yuan J, Wei J, Huang F, Wang F, Li G, Li Y, Xing L, Peng L, Yang M, Cao M, Zheng H, Wu W, Zou R, Li D, Xu Z, Wang H, Zhang M, Zhang Z, Gao GF, Jiang C, Liu L, Liu Y. Plasma IP-10 and MCP-3 levels are highly associated with disease severity and predict the progression of COVID-19. J Allergy Clin Immunol. 2020 Jul;146(1):119-127.e4. doi: 10.1016/j.jaci.2020.04.027. Epub 2020 Apr 29. PMID 32360286
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Marchandot B, Sattler L, Jesel L, Matsushita K, Schini-Kerth V, Grunebaum L, Morel O. COVID-19 Related Coagulopathy: A Distinct Entity? J Clin Med. 2020 May 31;9(6):1651. doi: 10.3390/jcm9061651. PMID 32486469
- [Background] Liu J, Zheng X, Tong Q, Li W, Wang B, Sutter K, Trilling M, Lu M, Dittmer U, Yang D. Overlapping and discrete aspects of the pathology and pathogenesis of the emerging human pathogenic coronaviruses SARS-CoV, MERS-CoV, and 2019-nCoV. J Med Virol. 2020 May;92(5):491-494. doi: 10.1002/jmv.25709. Epub 2020 Feb 21. PMID 32056249
- [Background] Panigrahy D, Gilligan MM, Huang S, Gartung A, Cortes-Puch I, Sime PJ, Phipps RP, Serhan CN, Hammock BD. Inflammation resolution: a dual-pronged approach to averting cytokine storms in COVID-19? Cancer Metastasis Rev. 2020 Jun;39(2):337-340. doi: 10.1007/s10555-020-09889-4. PMID 32385712
- [Background] Jentsch TJ, Stein V, Weinreich F, Zdebik AA. Molecular structure and physiological function of chloride channels. Physiol Rev. 2002 Apr;82(2):503-68. doi: 10.1152/physrev.00029.2001. PMID 11917096
- [Background] Petrat F, Boengler K, Schulz R, de Groot H. Glycine, a simple physiological compound protecting by yet puzzling mechanism(s) against ischaemia-reperfusion injury: current knowledge. Br J Pharmacol. 2012 Apr;165(7):2059-72. doi: 10.1111/j.1476-5381.2011.01711.x. PMID 22044190
- [Background] Weinberg JM, Bienholz A, Venkatachalam MA. The role of glycine in regulated cell death. Cell Mol Life Sci. 2016 Jun;73(11-12):2285-308. doi: 10.1007/s00018-016-2201-6. Epub 2016 Apr 11. PMID 27066896
- [Background] Zhong Z, Wheeler MD, Li X, Froh M, Schemmer P, Yin M, Bunzendaul H, Bradford B, Lemasters JJ. L-Glycine: a novel antiinflammatory, immunomodulatory, and cytoprotective agent. Curr Opin Clin Nutr Metab Care. 2003 Mar;6(2):229-40. doi: 10.1097/00075197-200303000-00013. PMID 12589194
- [Background] Gomez-Zamudio JH, Garcia-Macedo R, Lazaro-Suarez M, Ibarra-Barajas M, Kumate J, Cruz M. Vascular endothelial function is improved by oral glycine treatment in aged rats. Can J Physiol Pharmacol. 2015 Jun;93(6):465-73. doi: 10.1139/cjpp-2014-0393. Epub 2015 Mar 4. PMID 25988540
- [Background] Schemmer P, Zhong Z, Galli U, Wheeler MD, Xiangli L, Bradford BU, Conzelmann LO, Forman D, Boyer J, Thurman RG. Glycine reduces platelet aggregation. Amino Acids. 2013 Mar;44(3):925-31. doi: 10.1007/s00726-012-1422-8. Epub 2012 Nov 8. PMID 23135224
- [Background] Ikejima K, Iimuro Y, Forman DT, Thurman RG. A diet containing glycine improves survival in endotoxin shock in the rat. Am J Physiol. 1996 Jul;271(1 Pt 1):G97-103. doi: 10.1152/ajpgi.1996.271.1.G97. PMID 8760112
- [Background] Wheeler MD, Rose ML, Yamashima S, Enomoto N, Seabra V, Madren J, Thurman RG. Dietary glycine blunts lung inflammatory cell influx following acute endotoxin. Am J Physiol Lung Cell Mol Physiol. 2000 Aug;279(2):L390-8. doi: 10.1152/ajplung.2000.279.2.L390. PMID 10926563
- [Background] Iijima S, Shou J, Naama H, Calvano SE, Daly JM. Beneficial effect of enteral glycine in intestinal ischemia/reperfusion injury. J Gastrointest Surg. 1997 Jan-Feb;1(1):61-7; discussion 67-8. doi: 10.1007/s11605-006-0011-0. PMID 9834470
- [Background] Omasa M, Fukuse T, Toyokuni S, Mizutani Y, Yoshida H, Ikeyama K, Hasegawa S, Wada H. Glycine ameliorates lung reperfusion injury after cold preservation in an ex vivo rat lung model. Transplantation. 2003 Mar 15;75(5):591-8. doi: 10.1097/01.TP.0000053200.98125.14. PMID 12640295
- [Background] Alarcon-Aguilar FJ, Almanza-Perez J, Blancas G, Angeles S, Garcia-Macedo R, Roman R, Cruz M. Glycine regulates the production of pro-inflammatory cytokines in lean and monosodium glutamate-obese mice. Eur J Pharmacol. 2008 Dec 3;599(1-3):152-8. doi: 10.1016/j.ejphar.2008.09.047. Epub 2008 Oct 9. PMID 18930730
- [Background] Almanza-Perez JC, Alarcon-Aguilar FJ, Blancas-Flores G, Campos-Sepulveda AE, Roman-Ramos R, Garcia-Macedo R, Cruz M. Glycine regulates inflammatory markers modifying the energetic balance through PPAR and UCP-2. Biomed Pharmacother. 2010 Oct;64(8):534-40. doi: 10.1016/j.biopha.2009.04.047. Epub 2009 Oct 17. PMID 19864106
- [Background] Garcia-Macedo R, Sanchez-Munoz F, Almanza-Perez JC, Duran-Reyes G, Alarcon-Aguilar F, Cruz M. Glycine increases mRNA adiponectin and diminishes pro-inflammatory adipokines expression in 3T3-L1 cells. Eur J Pharmacol. 2008 Jun 10;587(1-3):317-21. doi: 10.1016/j.ejphar.2008.03.051. Epub 2008 Apr 8. PMID 18499099
- [Background] Wheeler MD, Thurman RG. Production of superoxide and TNF-alpha from alveolar macrophages is blunted by glycine. Am J Physiol. 1999 Nov;277(5):L952-9. doi: 10.1152/ajplung.1999.277.5.L952. PMID 10564180
- [Background] Anonimous. New and nonofficial remedies. J Am Med Assoc 1935;104:1241
- [Background] File SE, Fluck E, Fernandes C. Beneficial effects of glycine (bioglycin) on memory and attention in young and middle-aged adults. J Clin Psychopharmacol. 1999 Dec;19(6):506-12. doi: 10.1097/00004714-199912000-00004. PMID 10587285
- [Background] Fries MH, Rinaldo P, Schmidt-Sommerfeld E, Jurecki E, Packman S. Isovaleric acidemia: response to a leucine load after three weeks of supplementation with glycine, L-carnitine, and combined glycine-carnitine therapy. J Pediatr. 1996 Sep;129(3):449-52. doi: 10.1016/s0022-3476(96)70081-1. PMID 8804338
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Horowitz A, Kelly D. Double-blind, placebo-controlled, crossover trial of glycine adjuvant therapy for treatment-resistant schizophrenia. Br J Psychiatry. 1996 Nov;169(5):610-7. doi: 10.1192/bjp.169.5.610. PMID 8932891
- [Background] Heresco-Levy U, Javitt DC, Ermilov M, Mordel C, Silipo G, Lichtenstein M. Efficacy of high-dose glycine in the treatment of enduring negative symptoms of schizophrenia. Arch Gen Psychiatry. 1999 Jan;56(1):29-36. doi: 10.1001/archpsyc.56.1.29. PMID 9892253
- [Background] Khan M, Ron Van Der Wieken L, Riezebos RK, Tijssen JG, Kiemeneij F, Slagboom T, Laarman GJ. Oral administration of glycine in the prevention of restenosis after coronary angioplasty. A double blind placebo controlled randomized feasibility trial evaluating safety and efficacy of glycine in the prevention of restenosis after angioplasty. Acute Card Care. 2006;8(1):58-64. doi: 10.1080/14628840600643383. PMID 16720430
- [Background] Carvajal, G., et al., Inhibición de la glicosilación no enzimática de la hemoglobina en la diabetes mellitus. Rev Inst Nal Enf Resp 1995;8:185-188.
- [Background] Cruz M, Maldonado-Bernal C, Mondragon-Gonzalez R, Sanchez-Barrera R, Wacher NH, Carvajal-Sandoval G, Kumate J. Glycine treatment decreases proinflammatory cytokines and increases interferon-gamma in patients with type 2 diabetes. J Endocrinol Invest. 2008 Aug;31(8):694-9. doi: 10.1007/BF03346417. PMID 18852529
- [Background] Vargas MH, Del-Razo-Rodriguez R, Lopez-Garcia A, Lezana-Fernandez JL, Chavez J, Furuya MEY, Marin-Santana JC. Effect of oral glycine on the clinical, spirometric and inflammatory status in subjects with cystic fibrosis: a pilot randomized trial. BMC Pulm Med. 2017 Dec 15;17(1):206. doi: 10.1186/s12890-017-0528-x. PMID 29246256
- [Derived] Vargas MH, Chavez J, Del-Razo-Rodriguez R, Munoz-Perea C, Romo-Dominguez KJ, Baez-Saldana R, Rumbo-Nava U, Guerrero-Zuniga S. Lower Serum Magnesium Is Associated with Mortality in Severe COVID-19: A Secondary Analysis of a Randomized Trial. Biol Trace Elem Res. 2025 Nov;203(11):5987-5996. doi: 10.1007/s12011-025-04619-9. Epub 2025 Apr 15. PMID 40234280
- [Derived] Vargas MH, Chavez J, Del-Razo-Rodriguez R, Munoz-Perea C, Romo-Dominguez KJ, Baez-Saldana R, Rumbo-Nava U, Guerrero-Zuniga S. Glycine by enteral route does not improve major clinical outcomes in severe COVID-19: a randomized clinical pilot trial. Sci Rep. 2024 May 21;14(1):11566. doi: 10.1038/s41598-024-62321-7. PMID 38773199